CLINICAL TRIAL: NCT00000783
Title: Heterosexual HIV Transmission Study (HATS)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: HATS COUPLES
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Healthy
Keywords: Sex Behavior; Sexual Partners
MeSH Terms: conditions — HIV Infections; Sexual Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Seminal and cervico-vaginal fluids will be collected as well as blood and urine samples.

GROUPS / COHORTS (2):
- 1: Sexually active HIV-infected concordant couples
- 2: Sexually active HIV-infected discordant couples

SUMMARY:
PRIMARY: To identify sexual behaviors and biological factors associated with an increased risk of heterosexual HIV transmission.

SECONDARY: To assess the effect of safer sex counseling on behavior of sexually active heterosexuals in which one member of the couple is infected with HIV. To create a repository of serum, peripheral blood mononuclear cells, semen, and cervico-vaginal washings from heterosexual couples who are concordant (both partners HIV infected) and discordant (one partner HIV infected) with respect to HIV infection.

In the United States, the number of AIDS cases attributed to heterosexual transmission, although still a small percentage of the total number of reported cases, is the most rapidly growing category. The rate at which HIV is transmitted between heterosexual couples and the factors that may impede or enhance heterosexual transmission are important to understanding and slowing the worldwide HIV epidemic.

DETAILED DESCRIPTION:
In the United States, the number of AIDS cases attributed to heterosexual transmission, although still a small percentage of the total number of reported cases, is the most rapidly growing category. The rate at which HIV is transmitted between heterosexual couples and the factors that may impede or enhance heterosexual transmission are important to understanding and slowing the worldwide HIV epidemic.

This epidemiologic study is composed of three parts. PART A: In a prospective study, heterosexual couples who are discordant with respect to HIV infection will be evaluated at 6-month intervals to determine whether HIV transmission has occurred and to identify biological and behavioral factors associated with HIV transmission from the infected partner to the uninfected partner.

PART B: A case-control study will compare behavioral and biological data from heterosexual couples who are concordant for HIV infection at study entry with data from appropriate discordant couples enrolled in the prospective study. "Cases" will be HIV-infected secondary partners (from concordant couples) and "controls" will be uninfected secondary partners (from discordant couples).

PART C: In a cross-sectional study, semen and cervico-vaginal washings will be collected from HIV-infected men and women in Parts A and B and evaluated for presence of HIV by virologic and serologic methods.

Members of each couple will be interviewed separately by different interviewers. Demographic, sexual behavior and drug use history, and psychosocial information will be obtained. Participants will undergo clinical examination and various diagnostic laboratory tests (e.g., blood tests, urine screening, and gynecological tests). They will receive post-test counseling.

ELIGIBILITY:
Inclusion Criteria

Risk Behavior:

PART B ONLY:

* HIV-infected partner (primary partner) must have a known risk factor for HIV infection, such as
* Bisexual male.
* IV drug user.
* Hemophiliac male.
* Recipient of HIV-contaminated transfusion.

Participants must meet the following criteria:

* Heterosexual couples in which at least one member is HIV-infected. Comparison group consists of heterosexual couples concordant that are both HIV infected.
* Able to speak English or Spanish.

PART A secondary partners:

* Risk factor for HIV infection other than heterosexual contact, such as
* Evidence of any past or present parenteral drug use by self report, physical examination, or urine test.
* History of homosexual activity (if male) within 5 years prior to study entry.

PART B secondary partners:

* Risk factor for HIV infection other than sexual contact with the primary partner, such as
* Evidence of any past or present parenteral drug use by self-report or by urine test.
* History of homosexual activity (if male) at any time since 1978.
* Sexual contact with another person with an HIV risk factor at any time since 1978, unless secondary partner is documented to be HIV uninfected subsequent to the last contact with such person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sexually active HIV-infected concordant and discordant couples
Sampling Method: Non-Probability Sample
Dates: Start 1994-06; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
To identify sexual behaviors and biological factors associated with an increased risk of heterosexual HIV transmission | Throughout study

SECONDARY OUTCOMES:
To assess the effect of safer sex counseling on the behavior of sexually active heterosexuals in which one member of the couple is infected with HIV | Throughout study
To create a repository of serum, peripheral blood mononuclear cells, semen, and cervico-vaginal washings from heterosexual couples who are concordant (both partners HIV positive) and discordant (one partner HIV positive) with respect to HIV infection | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: O'Brien, Study Chair; Cordell, Study Chair
Locations (1):
- UMDNJ - New Jersey Med School, Newark, New Jersey, United States

REFERENCES:
- [Background] Cornell RG, Bromberg J, Grijalva K, Kelly P, Cordell J. Effects of changing recruitment patterns on risk factor estimates: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C324 (abstract no PoC 4477)
- [Background] Strug D, Des Jarlais D, Sogolow E, Handte J, Bromberg J, Cornell R, Cordell J, Landesman S. Types of sexual partner relationships and condom use among women in Brooklyn: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1991 Jun 16-21;7(2):324 (abstract no WC3112)
- [Background] Padian N, Bromberg J, O'Brien T, Vranizan K, Cordell J, Louria D, Van-Devanter N, Landesman S. Smoking and bleeding from trauma during sex: risks for heterosexual transmission of HIV. The HATS/CDC Research Group. Int Conf AIDS. 1993 Jun 6-11;9(2):648 (abstract no PO-C02-2588)
- [Background] Sogolow ED, Des Jarlais D, Landesman SH, Kelly P, Sampson-Lee G, Cordell J, Cornell R. The experience of participating in a cohort study of HIV transmission: a report from The Heterosexual HIV Transmission Study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(3):189 (abstract no PuC 8216)
- [Background] Bromberg J, Maher J, Wang W, Grijalva K, Cordell J. Within couple disagreement on condom use: a report from the heterosexual HIV transmission study (HATS/CDC). Int Conf AIDS. 1993 Jun 6-11;9(2):774 (abstract no PO-C33-3345)
- [Background] Wan J, Bromberg J, Cornell RG, Skurnick J, Cordell J, Vermund S. Generalized additive models for paired covariates in an HIV discordant couples study: a report from The Heterosexual HIV Transmission Study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(3):193 (abstract no PuC 8243)
- [Background] Bromberg J, Wan J, Cornell RG, Grijalva K, Cordell J, Kelly P, Landesman S. Entry criteria bias in studies of high-risk individuals: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C371 (abstract no PoC 4773)
- [Background] Skurnick J, Bromberg J, Cordell J, Foley M, Wang W, Louria D. Change in couples' sexual activity after knowledge of HIV discordance: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1992 Jul 19-24;8(2):C273 (abstract no PoC 4170)
- [Background] Skurnick J, Bromberg J, Grijalva K, Cordell J, Louria D, Monto A, Weiss S. Behavior changes in heterosexual couples discordant for HIV: a report from the heterosexual HIV transmission study (HATS). Int Conf AIDS. 1991 Jun 16-21;7(2):319 (abstract no WC3094)